CLINICAL TRIAL: NCT07234877
Title: A Randomized Phase II Study Evaluating Upfront SRT to All Brain Metastases Followed by Ivonescimab Plus Chemotherapy Versus Upfront Ivonescimab Plus Chemotherapy in Patients With Asymptomatic Active Brain Metastases From NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Summit Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 2456-LCG-BTG
Record Dates: First submitted 2025-09-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Ivonescimab; Phase II study
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequencing arm (Experimental): Patients will receive SRS/FSRT for all BM within ≤14 days from randomization, followed by 4 cycles of platinum-based chemotherapy combined with ivonescimab at 20 mg/kg every 3 weeks (Q3W). The systemic therapy will be followed by maintenance therapy with ivonescimab at 20 mg/kg plus pemetrexed (for patients with non-squamous NSCLC only) Q3W, for up to 2 years.
  Interventions: Drug: ivonescimab
- Systemic treatment alone arm (Experimental): Patients will receive 4 cycles of platinum-based chemotherapy combined with ivonescimab 20 mg/kg Q3W, followed by maintenance ivonescimab 20 mg/kg with pemetrexed (pemetrexed non-squamous only) Q3W for a maximum of 2 years.
  Interventions: Drug: ivonescimab

INTERVENTIONS:
Drug: ivonescimab — ivonescimab iv at 20 mg/kg every 3 weeks

SUMMARY:
This is a randomized, two-arm, comparative Phase II clinical trial designed to evaluate the difference in intracranial progression-free survival (iPFS) between two treatment strategies, assessed locally.

Approximately 158 patients will be randomized in a 1:1 ratio. Will be included patients with pathology proven metastatic NSCLC without an actionable genomic alteration for which there is first line targeted treatment available and active asymptomatic brain metastasis (newly diagnosed or progressive).

The primary objective is to compare iPFS between the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* ECOG PS <= 2
* Patients with pathology proven metastatic NSCLC without an actionable genomic alteration for which there is first line targeted treatment approved by EMA and recommended by the ESMO guidelines.
* Asymptomatic or clinically symptomatic brain metastases defined as requiring a dose of steroids of maximum 4 mg equivalent dexamethasone per day for the last 7 days to control neurological symptoms. With the clinically oligosymptomatic further defined as having no indication for immediate localized brain therapy, including neurosurgery or radiotherapy. Patients with controlled seizures can be enrolled.
* Newly diagnosed brain metastasis with the following characteristics:

  * 1-10 newly diagnosed and untreated (except resected) brain metastases Note: if the neuronavigation MRI in the upfront SRS/FSRT arms shows > 10 metastases, but the MRI used for enrolment showed 1-10 metastases, the patient will be still considered eligible.
  * At least one metastasis should be at least 5x5 mm. In case of doubt on the diagnosis of brain metastasis, the lesion should not be irradiated but followed up.
  * The largest metastasis must be <10 mL in volume and <30 mm in longest diameter (resected lesions would not count).
  * The maximum cumulative volume of brain metastases must be <30 mL (resected lesions would not count)
* Adequate Organ Function

Exclusion Criteria:

* Patients with oligometastatic NSCLC who are scheduled to receive radical local treatment to extra-cranial sites.
* Patients with contra-indications to brain MRI with gadolinium-based contrast agent.
* Active auto-immune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Patients with >30 Gy of chest radiation therapy within 6 months prior to randomization; non-thoracic radiation therapy >30Gy within 4 weeks prior to randomization, or palliative radiation therapy of ≤30 Gy within 7 days prior to randomization.
* Prior brain irradiation (including whole brain radiotherapy and SRS).
* Prior systemic treatment for metastatic NSCLC. Patients having received adjuvant or neoadjuvant chemotherapy or curative-intent chemoradiotherapy with or without PD-1/L1 inhibitors can be enrolled if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the development of metastatic disease.
* Major surgical procedures or serious trauma within 4 weeks prior to randomization or plans for major surgical procedures within 4 weeks after the first dose (as determined by the investigator). Minor local procedures (excluding central venous catheterization and port implantation) within 3 days prior to randomization.
* History of coagulopathy and/or clinically significant bleeding symptoms or risk within 4 weeks prior to randomization
* Poorly controlled hypertension with repeated systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg after oral antihypertensive therapy
* History of serious cardiovascular, gastronintestinal, thromboembolic, neurological, or pulmonary conditions before randomization.
* History of perforation of the gastrointestinal tract and/or fistula, history of gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive bowel resection (partial colectomy or extensive small bowel resection) within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-10 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression-free survival based on local assessment using RANO-BM criteria | First at week 6 and week 12 (±1 week) post-randomization. Then every 12 weeks (±2 weeks) until intracranial progression or study discontinuation.
  Time interval between the date of randomization and the date of intracranial progression or neurological related death, whichever occurs first

SECONDARY OUTCOMES:
Overall survival | Overall survival is defined as the time interval between the date of randomization and the date of death from any cause, assessed up to 4 years
Intracranial PFS as per central review | Intracranial PFS based on central assessment is defined as the time interval between the date of randomization and the date of intracranial progression or neurological related death, whichever occurs first, assessed up to 2 years
Intracranial overall response rate (icORR), based on RANO-BM criteria as per local assessment | The overall icORR is defined as the time interval between the date of randomization and the date of intracranial response, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lizza Hendriks, MD, PhD, Principal Investigator — Maastricht UMC